CLINICAL TRIAL: NCT02716714
Title: A Multi-center, OPen, InvEstigator Initiated Phase IV Clinical TRial to Evaluate the Efficacy and SaFety of Ingenol Mebutate Gel 0.015% on Face and Scalp & 0.05% on Trunk and Extremities in KorEan Patient With ACtinic KeraTosis (PERFECT)
Brief Title: Clinical Trial of Ingenol Mebutate Gel 0.015% & 0.05% in Actinic Keratosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University (Other)
Collaborators: LEO Pharma (Industry); Chonnam National University Hospital (Other); Severance Hospital (Other); Ajou University School of Medicine (Other); Asan Medical Center (Other); Samsung Medical Center (Other); Seoul National University Bundang Hospital (Other); Dong-A University Hospital (Other); Korea University Anam Hospital (Other); Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Il-Hwan Kim, Professor, Korea University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSSCLK2014-01
Record Dates: First submitted 2016-01-28; First posted 2016-03-23 (Estimated); Results first posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Actinic Keratosis
Keywords: Korean
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ingenol mebutate gel 0.015% (Active Comparator): Applied on face and scalp for three days.
  Interventions: Drug: ingenol mebutate gel 0.015%
- ingenol mebutate gel 0.05% (Active Comparator): Applied on trunk and extremities for two days.
  Interventions: Drug: ingenol mebutate gel 0.05%

INTERVENTIONS:
Drug: ingenol mebutate gel 0.015% — -Face or Scalp arm (Referred to Face/Scalp arm): Apply ingenol mebutate gel 0.015% once daily for 3 consecutive days
  Other Names: Picato® gel
  Arms: ingenol mebutate gel 0.015%
Drug: ingenol mebutate gel 0.05% — -Trunk or Extremities arm (Referred to Trunk/Extremities arm): Apply ingenol mebutate gel 0.05% once daily for 2 consecutive days
  Other Names: Picato® gel
  Arms: ingenol mebutate gel 0.05%

SUMMARY:
This study evaluate the efficacy and safety of ingenol mebutate gel 0.015% on face and scalp & 0.05% on trunk and extremities in Korean patient with actinic keratosis.

DETAILED DESCRIPTION:
The mechanism of action of ingenol mebutate for actinic keratosis(AK) treatment involves a rapid induction of necrosis followed by neutrophil-mediated, antibody-dependent cellular cytotoxicity (ADCC) of residual lesion. As the ingenol mebutate infiltrates the cell membrane, it increases intracellular Ca2+ concentration which leads to mitochondrial swelling and disruption of mitochondrial membrane within hours. The release of intra-mitochondrial Ca2+ into the cytoplasm leads to depletion of adenosine triphosphate (ATP) and a rapid induction of cell death by necrosis. This process occurs within 1 hour of application, which explains why the treatment period requires only 2 or 3 days of treatment. As the next phase, the cellular necrosis is accompanied by a robust inflammatory response through the release of proinflammatory cytokines from skin cells and tumor cells undergoing necrosis. The release of these proinflammatory cytokines into the dysplastic cells mediates the process of neutrophil recruitment through paracrine signaling and activation of endothelial cells. Here, the neutrophil mediated ADCC occurs, where activated neutrophils attach to the fragment, crystallized (Fc) parts of antibodies of dysplastic cells and destroys the residual dysplastic epidermal cells. In this way, the ingenol mebutate eradicates any residual tumor cells and prevents recurrence of actinic keratosis.As described above, the rapid effect and dual mechanism of action of ingenol mebutate gel allows not only a short-course therapy (2 or 3 days of application) for the elimination of actinic keratosis but also, the benefit for eradication of any residual lesions preventing the recurrence and the progression of AK into squamous cell carcinoma (SCC).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 19 years
2. Histopathologically diagnosed AK patients with at least 1 macroscopic and discrete lesion within a contiguous 25 cm2 (e.g. 5 cm x 5 cm) of treatment area
3. The treatment area including the lesion must be accessible to apply the investigational product. However, the lesions on lips, mucosa, outer ear (concha) and those around eyes are excluded.
4. Subjects who signed the written informed consent prior to perform any study-related procedures or assessments, including photographs of their treatment area for documentation and efficacy assessment.

Exclusion Criteria:

1. Hypersensitivity to any components of the investigational product
2. History or evidence of skin conditions that could interfere with evaluation of the investigational product(e.g., eczema, unstable psoriasis, xeroderma pigmentosa, inflammatory or infectious disease around the selected treatment area)
3. Unhealed wound within 5 cm, or basal cell carcinoma or squamous cell carcinoma within 10 cm from the selected treatment area.
4. Subjects who received or expected to receive any of the following pharmacotherapy and non-pharmacotherapy or procedures during the treatment and follow-up period
5. Subjects who have following disorder or abnormal laboratory result
6. Pregnant, lactating, and childbearing potential women who are unwilling to practice effective contraception; for example, oral contraceptives, hormonal methods, placement of an intrauterine device (IUD) or intrauterine system (IUS), barrier methods (i.e., condom or occlusive cap with spermicidal foam/gel/film/cream/suppository), male sterilization, and abstinence.
7. Subjects who previously underwent another clinical trial within 30 days or 5-times the half-life of previous investigational product prior to baseline (the longer period of time must be considered).
8. Other conditions by investigator's discretion to be inappropriate for this clinical study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilhwan Kim, MD, Principal Investigator — Korea University Ansan Hospital
Locations (1):
- Korea University Ansan Hospital, Ansan-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made within 6months of study completion.

REFERENCES:
- [Result] Callen JP, Bickers DR, Moy RL. Actinic keratoses. J Am Acad Dermatol. 1997 Apr;36(4):650-3. doi: 10.1016/s0190-9622(97)70265-2. No abstract available. PMID 9092763
- [Result] Schmitt JV, Miot HA. Actinic keratosis: a clinical and epidemiological revision. An Bras Dermatol. 2012 May-Jun;87(3):425-34. doi: 10.1590/s0365-05962012000300012. PMID 22714759
- [Result] Brash DE, Ziegler A, Jonason AS, Simon JA, Kunala S, Leffell DJ. Sunlight and sunburn in human skin cancer: p53, apoptosis, and tumor promotion. J Investig Dermatol Symp Proc. 1996 Apr;1(2):136-42. PMID 9627707
- [Result] Flohil SC, van der Leest RJ, Dowlatshahi EA, Hofman A, de Vries E, Nijsten T. Prevalence of actinic keratosis and its risk factors in the general population: the Rotterdam Study. J Invest Dermatol. 2013 Aug;133(8):1971-8. doi: 10.1038/jid.2013.134. Epub 2013 Mar 19. PMID 23510990
- [Result] Rossi R, Mori M, Lotti T. Actinic keratosis. Int J Dermatol. 2007 Sep;46(9):895-904. doi: 10.1111/j.1365-4632.2007.03166.x. No abstract available. PMID 17822489
- [Result] Salasche SJ. Epidemiology of actinic keratoses and squamous cell carcinoma. J Am Acad Dermatol. 2000 Jan;42(1 Pt 2):4-7. doi: 10.1067/mjd.2000.103342. PMID 10607349
- [Result] Kim HS, Cho EA, Bae JM, Yu DS, Oh ST, Kang H, Park CJ, Lee JD, Lee JY, Kim SY, Kim HO, Park YM. Recent trend in the incidence of premalignant and malignant skin lesions in Korea between 1991 and 2006. J Korean Med Sci. 2010 Jun;25(6):924-9. doi: 10.3346/jkms.2010.25.6.924. Epub 2010 May 24. PMID 20514316
- [Result] Slaper H, Velders GJ, Daniel JS, de Gruijl FR, van der Leun JC. Estimates of ozone depletion and skin cancer incidence to examine the Vienna Convention achievements. Nature. 1996 Nov 21;384(6606):256-8. doi: 10.1038/384256a0. PMID 8918873
- [Result] Nelson CG. Diclofenac gel in the treatment of actinic keratoses. Ther Clin Risk Manag. 2011;7:207-11. doi: 10.2147/TCRM.S12498. Epub 2011 Jun 15. PMID 21753882
- [Result] Stockfleth E, Ferrandiz C, Grob JJ, Leigh I, Pehamberger H, Kerl H; European Skin Academy. Development of a treatment algorithm for actinic keratoses: a European Consensus. Eur J Dermatol. 2008 Nov-Dec;18(6):651-9. doi: 10.1684/ejd.2008.0514. Epub 2008 Oct 27. PMID 18955209
- [Result] Anderson L, Schmieder GJ, Werschler WP, Tschen EH, Ling MR, Stough DB, Katsamas J. Randomized, double-blind, double-dummy, vehicle-controlled study of ingenol mebutate gel 0.025% and 0.05% for actinic keratosis. J Am Acad Dermatol. 2009 Jun;60(6):934-43. doi: 10.1016/j.jaad.2009.01.008. PMID 19467365
- [Result] Vegter S, Tolley K. A network meta-analysis of the relative efficacy of treatments for actinic keratosis of the face or scalp in Europe. PLoS One. 2014 Jun 3;9(6):e96829. doi: 10.1371/journal.pone.0096829. eCollection 2014. PMID 24892649
- [Result] Lebwohl M, Dinehart S, Whiting D, Lee PK, Tawfik N, Jorizzo J, Lee JH, Fox TL. Imiquimod 5% cream for the treatment of actinic keratosis: results from two phase III, randomized, double-blind, parallel group, vehicle-controlled trials. J Am Acad Dermatol. 2004 May;50(5):714-21. doi: 10.1016/j.jaad.2003.12.010. PMID 15097955
- [Result] Rosen RH, Gupta AK, Tyring SK. Dual mechanism of action of ingenol mebutate gel for topical treatment of actinic keratoses: rapid lesion necrosis followed by lesion-specific immune response. J Am Acad Dermatol. 2012 Mar;66(3):486-93. doi: 10.1016/j.jaad.2010.12.038. Epub 2011 Nov 4. PMID 22055282
- [Result] Lebwohl M, Swanson N, Anderson LL, Melgaard A, Xu Z, Berman B. Ingenol mebutate gel for actinic keratosis. N Engl J Med. 2012 Mar 15;366(11):1010-9. doi: 10.1056/NEJMoa1111170. PMID 22417254
- [Result] Lebwohl M, Shumack S, Stein Gold L, Melgaard A, Larsson T, Tyring SK. Long-term follow-up study of ingenol mebutate gel for the treatment of actinic keratoses. JAMA Dermatol. 2013 Jun;149(6):666-70. doi: 10.1001/jamadermatol.2013.2766. PMID 23553119
- See also: National Institute for Clinical Excellence. Guidance on Cancer Services:Improving outcomes for people with skin tumours including melanoma. The manual. February 2006. — http://www.nice.org.uk/guidance/csgstim/resources/improving-outcomes-for-people-with-skin-tumoursincluding-melanoma-the-manual-2006-guidance2

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients with actinic keratosis (AK) patients with the lesions on the face, scalp, trunk and/or extremities from 10 academic medical centers in South Korea. First subject was enrolled on 06 Apr 2015 and Last subject was completed on 13 Jun 2016.
Groups:
- Ingenol Mebutate Gel 0.015%: Participants with actinic keratosis on the face or scalp received 1 tube of ingenol mebutate gel 0.015% to be self-applied to the selected treatment area once daily for 3 consecutive days.
  1 tube (0.47g) contained the amount that can be applied to the area of approximately 25cm2(eg. cn. 5cm X 5cm) and 1 tube was applied to the selected treatment area.
- Ingenol Mebutate Gel 0.05%: Participants with actinic keratosis on the trunk or extremities received 1 tube of ingenol mebutate gel 0.05% to be self-applied to the selected treatment area once daily for 2 consecutive days.
  1 tube (0.47g) contained the amount that can be applied to the area of approximately 25cm2(eg. cn. 5cm X 5cm) and 1 tube was applied to the selected treatment area.
Period: Overall Study
Arm/Group | Ingenol Mebutate Gel 0.015% | Ingenol Mebutate Gel 0.05%
Started | 67 | 10
Completed | 55 | 8
Not Completed | 12 | 2

BASELINE CHARACTERISTICS:
Population: Of 91 screened subjects, 77 subjects were enrolled and included in Safety Set (Face or Scalp Group: 67, Trunk or Extremities Group: 10). After excluding 4 subjects for missing primary efficacy assessment, 73 subjects (Face or Scalp Group: 64, Trunk or Extremities Group: 9) were included in ITT Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ingenol Mebutate Gel 0.015% | Ingenol Mebutate Gel 0.05% | Total
Number analyzed (Participants) | 64 | 9 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 73 participants of overall number of baseline participants are analyzed as Intention To Treat (ITT) set. Intention To Treat (ITT) set was defined as all subjects who applied the investigational product at least once after the enrollment and allocation during this study and conducted the assessment of the primary efficacy measure.
  years | 72.39 (8.85) | 72.11 (5.44) | 72.36 (8.47)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 73 participants of overall number of baseline participants are analyzed as Intention To Treat (ITT) set. Intention To Treat (ITT) set was defined as all subjects who applied the investigational product at least once after the enrollment and allocation during this study and conducted the assessment of the primary efficacy measure.
  Participants
    Female | 46 | 4 | 50
    Male | 18 | 5 | 23
Fitzpatrick skin type [Count of Participants; unit: Participants] — Fitzpatrick skin type was described as following; Type I: Extremely fair skin, always burns, never tans Type II: Fair skin, always burns, sometimes tans Type III: Medium skin, sometimes burns, always tans Type IV: Olive skin, rarely burns, always tans Type V: Moderately pigmented brown skin, never burns, always tans Type VI: Markedly pigmented black skin, never burns, always tans and it was considered worse outcomes from type IV upto type VI. Population: Intent to treat population(Intention To Treat (ITT) set was defined as all subjects who applied the investigational product at least once after the enrollment and allocation during this study).
  Participants
    I | 0 | 0 | 0
    II | 7 | 1 | 8
    III | 42 | 6 | 48
    IV | 15 | 2 | 17
    V | 0 | 0 | 0
    VI | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] — Population: Intent to treat population(all participants who applied the investigational product at least once after the enrollment and allocation during this study).
  cm | 157.64 (7.72) | 159.89 (5.75) | 157.92 (7.51)
Weight [Mean (Standard Deviation); unit: kg] — Population: Intent to treat population(all participants who applied the investigational product at least once after the enrollment and allocation during this study).
  kg | 56.42 (8.89) | 60.24 (8.98) | 56.89 (8.93)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: Intent to treat population(all participants who applied the investigational product at least once after the enrollment and allocation during this study).
  kg/m^2 | 22.62 (2.59) | 23.49 (2.63) | 22.73 (2.60)
Actinic keratosis duration [Mean (Standard Deviation); unit: months] — Population: Intent to treat population(all participants who applied the investigational product at least once after the enrollment and allocation during this study).
  months | 8.43 (26.73) | 19.10 (52.48) | 9.74 (30.72)
Actinic keratosis duration at the selected treatment area [Mean (Standard Deviation); unit: months] — Population: Intent to treat population(all participants who applied the investigational product at least once after the enrollment and allocation during this study).
  months | 2.03 (8.67) | 1.03 (1.78) | 1.91 (8.14)
Severity of actinic keratosis [Count of Participants; unit: Participants] — Population: Intent to treat population(all participants who applied the investigational product at least once after the enrollment and allocation during this study).
  Participants
    AK I (Mild) | 9 | 3 | 12
    AK II (Moderate) | 42 | 5 | 47
    AK III (Severe) | 13 | 1 | 14
Prior treatment history of actinic keratosis [Count of Participants; unit: Participants] — Population: Intent to treat population(all participants who applied the investigational product at least once after the enrollment and allocation during this study).
  Participants
    Yes | 12 | 3 | 15
    No | 52 | 6 | 58

OUTCOME MEASURES:

1. Primary Outcome: CC Rate of AK Lesions in the Selected Treatment Area
Description: Complete Clearance (CC) means that clearance of all visible AK lesions in the selected treatment area and Investigator-rated actinic keratiosis(AK) lesion complete clearance (CC) rate at the selected treatment area on day 57 was analyzed.
Time Frame: at day 57
Population: Intent to treat population(all participants who applied the investigational product at least once after the enrollment and allocation during this study).
Measure: Count of Participants; unit: Participants
Arm/Group | Ingenol Mebutate Gel 0.015% | Ingenol Mebutate Gel 0.05%
Number analyzed (Participants) | 64 | 9
Participants
  CC | 49 | 8
  Non-CC | 15 | 1

2. Secondary Outcome: Percentage Change of the Number of AK Lesions in the Selected Treatment Area
Description: Percentage change from baseline in the number of actinic keratiosis(AK) lesions in the selected treatment area on Day 57 was analyzed.
Time Frame: Baseline and Day 57
Population: Intent to treat population(Intention To Treat (ITT) set was defined as all subjects who applied the investigational product at least once after the enrollment and allocation during this study).
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Ingenol Mebutate Gel 0.015% | Ingenol Mebutate Gel 0.05%
Number analyzed (Participants) | 64 | 9
percentage change | -80.08 (38.36) | -88.89 (33.33)

3. Secondary Outcome: Sustained CC Rate in CC Group
Description: Sustained Complete Clearance means that Complete Clearance was maintained until Month 6 in complete clearance (CC) group and sustained complete clearance(CC) rate at month 6 for complete clearance(CC) group was analyzed.
Time Frame: at 6 months
Population: In intent to treat population(all participants who applied the investigational product at least once after the enrollment and allocation during this study), CC Group consisted of 54 participants who had at least 1 follow-up after achieving complete clearance of AK lesions on Day 57.
Measure: Count of Participants; unit: Participants
Arm/Group | Ingenol Mebutate Gel 0.015% | Ingenol Mebutate Gel 0.05%
Number analyzed (Participants) | 47 | 7
Participants
  Sustained CC | 42 | 6
  Recurrence | 5 | 1

4. Secondary Outcome: Recurrence Rate in CC Group
Description: Recurrence rate in complete clearance(CC) group was analyzed.
Time Frame: at 6 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Ingenol Mebutate Gel 0.015% | Ingenol Mebutate Gel 0.05%
Number analyzed (Participants) | 47 | 7
Participants
  Recurrence rate | 5 | 2
  Censored | 42 | 5

5. Secondary Outcome: Percentage Change of the Number of AK Lesions in the Selected Treatment Area of CC Group
Description: Percentage change from baseline in the number of actinic keratiosis(AK) lesions at Month 6 in the selected treatment area in complete clearance(CC) Group was analyzed.
Time Frame: at 6 months from baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Ingenol Mebutate Gel 0.015% | Ingenol Mebutate Gel 0.05%
Number analyzed (Participants) | 47 | 7
Percentage change | -88.65 (37.61) | -85.71 (37.80)

6. Secondary Outcome: Change From Baseline in Quality of Life (Skindex-29)
Description: Skindex-29 is a self-administered QoL questionnaire comprised of 29 items scored on a 5-point scale (0=never, 1=rarely, 2=sometimes, 3=often, 4=all the time) covering 3 domains: emotional (10 items), symptomatic (7 items), and functional (12 items), with domain scores ranging from 0 to 40, 28, and 48, respectively. Lower scores for each of the domains represents a better Quality of life.
Time Frame: at 29 and 57 days from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ingenol Mebutate Gel 0.015% | Ingenol Mebutate Gel 0.05%
Number analyzed (Participants) | 64 | 9
units on a scale
  Emotions(Baseline): number analyzed (Participants) | 61 | 9
  Emotions(Baseline) | 20.57 (20.62) | 27.22 (19.94)
  Emotions(Day 29): number analyzed (Participants) | 62 | 9
  Emotions(Day 29) | 21.21 (20.24) | 12.50 (11.59)
  Emotions(Day 57): number analyzed (Participants) | 63 | 9
  Emotions(Day 57) | 15.28 (19.18) | 12.78 (16.56)
  Emotions(Day 29-Baseline): number analyzed (Participants) | 59 | 9
  Emotions(Day 29-Baseline) | -0.42 (21.96) | -14.72 (20.17)
  Emotions(Day 57-Baseline): number analyzed (Participants) | 60 | 9
  Emotions(Day 57-Baseline) | -6.46 (18.62) | -14.44 (20.49)
  Symptoms(Baseline): number analyzed (Participants) | 61 | 9
  Symptoms(Baseline) | 16.45 (17.54) | 31.35 (18.45)
  Symptoms(Day 29): number analyzed (Participants) | 62 | 9
  Symptoms(Day 29) | 20.16 (17.52) | 13.89 (8.83)
  Symptoms(Day 57): number analyzed (Participants) | 63 | 9
  Symptoms(Day 57) | 12.41 (14.86) | 12.70 (14.19)
  Symptoms(Day 29-Baseline): number analyzed (Participants) | 59 | 9
  Symptoms(Day 29-Baseline) | 3.09 (22.15) | -17.46 (17.08)
  Symptoms(Day 57-Baseline): number analyzed (Participants) | 60 | 9
  Symptoms(Day 57-Baseline) | -4.76 (19.71) | -18.65 (19.62)
  Functioning(Baseline): number analyzed (Participants) | 61 | 9
  Functioning(Baseline) | 8.54 (13.64) | 13.43 (11.13)
  Functioning(Day 29): number analyzed (Participants) | 62 | 9
  Functioning(Day 29) | 17.10 (20.19) | 5.56 (7.29)
  Functioning(Day 57): number analyzed (Participants) | 63 | 9
  Functioning(Day 57) | 10.58 (16.97) | 3.24 (7.52)
  Functioning(Day 29-Baseline): number analyzed (Participants) | 59 | 9
  Functioning(Day 29-Baseline) | 8.02 (21.32) | -7.87 (14.08)
  Functioning(Day 57-Baseline): number analyzed (Participants) | 60 | 9
  Functioning(Day 57-Baseline) | 1.45 (15.60) | -10.19 (14.67)

7. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM)
Description: Participants personally completed the tool to evaluate satisfaction with drug treatment. It consisted of 4 areas of Effectiveness, side effect, convenience, and global satisfaction, with a total of 14 sub-items. The full mark is 100, and it is divided in four stages as follows.
  * Very good: 76 -100 score
  * Good: 51-75 score
  * Not bad: 26-50 score
  * Bad: 0-25 score Scores for each area ranged from 0 to 100, with higher scores indicating that fewer side effects had occurred and greater treatment satisfaction.
Time Frame: at 29 and 57 days from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ingenol Mebutate Gel 0.015% | Ingenol Mebutate Gel 0.05%
Number analyzed (Participants) | 64 | 9
units on a scale
  Effectiveness(Day 29): number analyzed (Participants) | 62 | 9
  Effectiveness(Day 29) | 57.62 (18.88) | 61.11 (11.79)
  Effectiveness(Day 57) | 62.67 (16.22) | 70.37 (14.70)
  Side-effect(Day 29): number analyzed (Participants) | 62 | 9
  Side-effect(Day 29) | 84.48 (22.40) | 91.67 (14.99)
  Side-effect(Day 57) | 89.26 (19.84) | 91.41 (21.89)
  Convenience(Day 29): number analyzed (Participants) | 62 | 9
  Convenience(Day 29) | 60.75 (17.38) | 61.11 (15.96)
  Convenience(Day 57) | 65.10 (15.85) | 65.43 (16.62)
  Global satisfaction(Day 29): number analyzed (Participants) | 62 | 9
  Global satisfaction(Day 29) | 59.22 (18.89) | 65.08 (14.48)
  Global satisfaction(Day 57) | 60.60 (18.27) | 63.49 (21.26)

8. Secondary Outcome: Cosmetic Outcomes Assessment (COA)
Description: The investigator rated the subject's Cosmetic Outcomes Assessment(COA) using 5 grades (Very good, Good, No change, Bad, Very bad), and results were as follows.
Time Frame: at 29 and 57 days from baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ingenol Mebutate Gel 0.015% | Ingenol Mebutate Gel 0.05%
Number analyzed (Participants) | 64 | 9
Participants
  Day 29: number analyzed (Participants) | 62 | 9
  Day 29: Very good | 16 | 3
  Day 29: Good | 33 | 4
  Day 29: No change | 5 | 1
  Day 29: Bad | 8 | 1
  Day 29: Very bad | 0 | 0
  Day 57: Very good | 17 | 4
  Day 57: Good | 39 | 5
  Day 57: No change | 6 | 0
  Day 57: Bad | 2 | 0
  Day 57: Very bad | 0 | 0

9. Secondary Outcome: Time to Relapse in CC Group
Description: Time to relapse in complete clearance(CC) Group was analyzed. Median survival time with 95% confidence interval was calculated by Kaplan-Meier method.
Time Frame: at 6 months
Population: CC Group consisted of 54 participants who had at least 1 follow-up after achieving Complete Clearance of AK lesions on Day 57.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ingenol Mebutate Gel 0.015% | Ingenol Mebutate Gel 0.05%
Number analyzed (Participants) | 47 | 7
days | NA [144.00 to NA] — It wasn't calculated due to a low Recurrence rate (95% Confidence Interval: [144.00, NA]). | 203 [129.00 to 203.00]

10. Other Pre Specified Outcome: Medication for Actinic Keratosis
Description: The count of participants in complete clearance(CC) group and Non-CC group who administered medication for actinic keratosis on the selected treatment area after Day 57 was collected.
Time Frame: from 57 days to 6 months
Population: The number of participants who had at least 1 follow-up after assessment of treatment response on Day 57 was 67 and which is consisit of CC group(54 participants) and Non-CC group(13 participants). The CC group and Non-CC group for Ingenol Mebutate Gel 0.015% and 0.05% were intended to be analyzed together.
Measure: Count of Participants; unit: Participants
Groups:
- CC Group: The participants who achieved complete clearance of AK lesions in the selected treatment.
- Non-CC Group: The participants who didn't achieved complete clearance of AK lesions in the selected treatment.
Arm/Group | CC Group | Non-CC Group
Number analyzed (Participants) | 54 | 13
Participants
  Fluorouracil | 0 | 1
  Imiquimod | 1 | 0

11. Other Pre Specified Outcome: Non-Drug Treatment/Surgery for Actinic Keratosis
Description: The count of participants in complete clearance(CC) group and Non-CC group who received non-drug treatment/surgery for actinic keratosis on the selected treatment area after Day 57 was collected.
Time Frame: from 57 days to 6 months
Population: The number of participants who had at least 1 follow-up after assessment of treatment response on Day 57 and which is consisit of CC group(54 participants) and Non-CC group(13 participants). The CC group /Non-CC group for Ingenol Mebutate Gel 0.015% and 0.05% were intended to be analyzed together.
Measure: Count of Participants; unit: Participants
Groups:
- CC Group: The participants who achieved complete clearance of AK lesions in the selected treatment and the CC group of Ingenol Mebutate Gel 0.015% and 0.05% was intended to be analyzed together.
- Non-CC Group: The participants who didn't achieved complete clearance of AK lesions in the selected treatment and the Non-CC group of Ingenol Mebutate Gel 0.015% and 0.05% was intended to be analyzed together.
Arm/Group | CC Group | Non-CC Group
Number analyzed (Participants) | 54 | 13
Participants
  Skin cryotherapy | 5 | 4
  Photodynamic therapy | 0 | 1
  Phototherapy | 0 | 1
  Skin lesion excision | 1 | 0
  Wound treatment | 1 | 0
  Biopsy skin | 0 | 1

ADVERSE EVENTS:
Arm/Group | Ingenol Mebutate Gel 0.015% | Ingenol Mebutate Gel 0.05%
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/67 | 0/10
Other Adverse Events (participants affected / at risk) | 67/67 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ingenol Mebutate Gel 0.015% (N=67) | Ingenol Mebutate Gel 0.05% (N=10)
Squamous cell carcinoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ingenol Mebutate Gel 0.015% (N=67) | Ingenol Mebutate Gel 0.05% (N=10)
Erythema (Skin and subcutaneous tissue disorders) | 65 | 9
Scab (Skin and subcutaneous tissue disorders) | 62 | 8
Skin exfoliation (Skin and subcutaneous tissue disorders) | 62 | 6
Blister (Skin and subcutaneous tissue disorders) | 55 | 7
Skin swelling (Skin and subcutaneous tissue disorders) | 51 | 5
Skin erosion (Skin and subcutaneous tissue disorders) | 49 | 4
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 6 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Administration site pain (General disorders) | 11 | 3
Swelling (General disorders) | 1 | 2
Rash pustular (Infections and infestations) | 7 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Folliculitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Tinea pedis (Infections and infestations) | 1 | 0
Ichthyosis (Congenital, familial and genetic disorders) | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes